| Official Title: Risk of Aspergillus infection in patients with chronic |
|---|
| structural lung disease |
| Short Title: Risk of Aspergillus infection in patients with chronic lung disease |
| NCT Number: Pending |
| Study Duration: July 1, 2022 - January 31, 2024 |
| Funding Source: Sichuan Provincial People's Hospital |
| Principal Investigator: Dr. Lin Chen |
| Affiliation: Sichuan Provincial People's Hospital |
| Address: 32# W. Sec 2, 1st Ring Rd., Chengdu, Sichuan, China |

**Contact Information:** 

Email: chenlinhx@med.uestc.edu.cn

Phone: +86 18111585286

**Document Date:** January 31, 2024

### **Informed Consent Form**

Research Project: Risk of Aspergillus infection in patients with chronic structural lung disease.

**Research Purpose:** This study aims to identify the risk factors associated with fungal infections and to investigate acute exacerbation in these patients.

# **Study Process:**

Participants will undergo the following procedures:

- Sputum Microscopy and Culture: To check for the presence of Aspergillus.
- High-Resolution Computed Tomography (HRCT) of the Chest: To obtain detailed images of the lung structure.
- Blood Tests: Including tests for Aspergillus-specific IgG and IgM antibodies and serum galactomannan (GM).

The data from patients diagnosed with Aspergillus infection will be compared to those with Aspergillus colonization to understand risk factors better.

### Possible Risks and Discomfort:

Participants may experience minor side effects during blood collection:

- <u>Pain</u>: Brief pain during needle insertion.
- <u>Bleeding</u>: Minor bleeding at the puncture site.

- <u>Infection</u>: Rare, as strict sterilization protocols are followed.
- Other unforeseeable situations: Any severe reaction will lead to immediate cessation of the procedure.

**Data Collection and Privacy:** All personal information will be confidential. Results will be anonymized to protect participant privacy.

**Voluntary Participation:** Participation is voluntary, and participants can withdraw at any time without affecting their medical care or rights.

## Follow-up Period and Benefits:

- <u>Free Diagnostic Testing</u>: Participants will receive free testing for Aspergillus-specific IgG and IgM antibodies, with each participant eligible for at least two free tests. Additional tests during the follow-up period may be requested by the overseeing physician based on treatment progress, at no cost to the participant.
  - Free Outpatient Follow-up Visits:
  - One-Month Follow-up: All participants will benefit from free follow-up visits at our outpatient clinic for one month after initial participation. These visits are designed to monitor health outcomes and provide ongoing support.
  - o Extended Six-Month Follow-up for Positive Cases: Participants who test positive for Aspergillus infection will receive an extended follow-up period of six months. During this time, they will continue to have free access to monthly outpatient follow-up visits, ensuring comprehensive monitoring and care throughout their treatment course.

#### **Consent Statement:**

(Project Leader: Lin Chen, 18111585286).

| I have read the above information, fully understood the study process, possible risks and discomforts, data collection, |
|---|
| and privacy protection. I voluntarily participate in this study and allow blood test data to be used for research |
| purposes. |
| Patient or Authorized Family Member's Signature: Date: |
| Conversing Doctor's Signature: Date: |
| *This study has been submitted to and approved by the Ethics Review Committee of Sichuan Provincial |
| People's Hospital, affiliated with Sichuan Academy of Medical Sciences (Approval No. Lun Audit (Research) |
| 2023-482). All study participants will undergo a detailed informed consent process to ensure they fully understand the |
| study's purpose, process, potential risks, and benefits, and are aware of their right to withdraw from the study at any |
| time. |
| If participants have any questions about this study, please feel free to contact the study team doctor |